CLINICAL TRIAL: NCT01641328
Title: Phase 1 Study of Cognitive Activation Behavioral Therapy for MCI: A Randomized Waitlist-Control and Delayed Active-Control Study
Brief Title: Cognitive Activation Therapy for MCI: A Randomized Control Study
Acronym: FarbMCI2012
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rotman Research Institute at Baycrest (Other)
Collaborators: Roy Hintsa (Unknown)
Responsible Party: Principal Investigator, Norman Farb, Postdoctoral Fellow, Rotman Research Institute at Baycrest
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RRI_Farb_001
Record Dates: First submitted 2012-07-12; First posted 2012-07-16 (Estimated); Last update posted 2012-07-16 (Estimated); Status verified 2012-07

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild Cognitive Impairment; MCI; Meditation; Mindfulness; Cognitive Activation; Cognitive Training; Tai Chi
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waitlist Control / Home-based training (Active Comparator): This group will serve as a waitlist control group while the active group is performing training. Following assessment at the end of the active group period, this group will begin home-based training and will be assessed at the end of that 10 week period.
  Interventions: Behavioral: Waitlist Control / Home-based training
- Cognitive Activation Group (Experimental): This group will attend the 3/week group intervention meetings over 10 weeks.
  Interventions: Behavioral: Cogntive Activation Training

INTERVENTIONS:
Behavioral: Cogntive Activation Training — Mindfulness-based stress reduction - 30 minutes / class x 3 classes / week; optional home practice Tai Chi - 30 minutes / class x 3 classes / week; optional home practice Computer-based cognitive training - 20 minutes / class x 3 classes / week; optional home practice
  Other Names: Computer-based cognitive training is provided by Lumosity
  Arms: Cognitive Activation Group
Behavioral: Waitlist Control / Home-based training — Computer-based cognitive training - 20 minutes / day Daily walking - 20 minutes / day Biofeedback relaxation Training - 20 minutes / day
  Other Names: Computer-based cognitive training is provided by Lumosity; Biofeedback relaxation training is provided by HeartMath
  Arms: Waitlist Control / Home-based training

SUMMARY:
Mild cognitive impairment (MCI) describes an initial phase of cognitive decline, usually among older adults, in which a person notices a decline in attention or memory, and performs worse than normal on cognitive tests of such. People with MCI are more likely to develop Alzheimer's disease or related dementia than others their same age, and so MCI is thought of as an early warning sign of progressive cognitive decline.

While some forms of MCI may be brought about by purely genetic causes, other cases may be due to a withdrawal of cognitive engagement with the world. In these cases, a rigorous program of cognitive training may be beneficial, halting or reversing symptom progression.

The current study will evaluate a multifaceted cognitive activation program on older adults with MCI. This group program is intensive, running for 10 weeks, 3 times per week, for a total of 100 hours of training. Training consists of meditation exercises for broad attention activation, Tai Chi exercises to integrate cognition with body awareness, and cognitive training through computerized attention, memory, and problem solving exercise.

Subjective impressions and objective measures of cognitive ability will be measured before and after the intervention. The investigators will also examine effects on mood and levels of daily function. Results will be compared to a waitlisted control group. The control group will subsequently be entered into a home-based version of the program for 10 weeks, with assessment before and after training, to look at the importance of the group meeting dynamic in promoting cognitive change.

ELIGIBILITY:
Inclusion Criteria:

* Subjective complaint about decline in memory or attention
* > 1 deviation below age-norm performance on memory or attention tasks
* Independence in daily living
* English speaking

Exclusion Criteria:

* Neurological disorders (including aphasias) or reversible causes of dementia (e.g., hypothyroidism or B12 deficiency)
* Montreal Cognitive Assessment (MOCA) score < 24
* Clinical mood disorder such as depression or anxiety
* Other serious medical conditions that preclude participation in the program

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-03 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Processing Speed | Before and After Intervention
  Processing speed on computerized cognitive task.
Memory | Before and After Intervention
  Tests of immediate recall and delayed recall, recognition, and familiarity.
Executive Function | Before and After Intervention
  Tests of inhibition, task switching, and problem solving.
Attention / Working Memory | Before and after intervention
  Working memory measures such as digit span, selection of targets among distractors, etc.

SECONDARY OUTCOMES:
Mood and Well-being | Before and after intervention
  Tests of dysphoric affect and subjective quality of life
Daily Function | Before and after intervention
  Tests of instrumental activities of daily living

CONTACTS AND LOCATIONS:
Locations (1):
- Baycrest, Toronto, Ontario, Canada

REFERENCES:
- See also: Related info about Baycrest and the Rotman Research Institute — http://research.baycrest.org/